CLINICAL TRIAL: NCT06935175
Title: A Study of SHR-1826 Monotherapy or in Combination With Immunotherapy in Patients With Advanced Hepatocellular Cancer
Brief Title: A Study of SHR-1826 Monotherapy or in Combination With Immunotherapy in the Treatment of Advanced Hepatocellular Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-2nd-IIT-SHR1826-SHR1316
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Cancer
Keywords: hepatocellular cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1826 monotherapy arm (Experimental)
  Interventions: Drug: SHR-1826
- SHR-1826 and immunotherapy combination therapy (Experimental)
  Interventions: Drug: SHR-1826 and immunotherapy combination therapy

INTERVENTIONS:
Drug: SHR-1826 — SHR-1826 will be administrated per dose level in which the patients are assigned.
  Arms: SHR-1826 monotherapy arm
Drug: SHR-1826 and immunotherapy combination therapy — SHR-1826 and immunotherapy will be administrated per dose level in which the patients are assigned.
  Arms: SHR-1826 and immunotherapy combination therapy

SUMMARY:
The study was designed to evaluate the efficacy and safety of SHR-1826 monotherapy or in combination with immunotherapy in the treatment of advanced hepatocellular cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1.18-75 years old, male or female.

2.Hepatocellular carcinoma diagnosed histologically or cytologically, and not suitable for radical surgery;

3.Failure of at least one line of standard treatment (progression or intolerance);

4.According to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1), there is at least one measurable lesion diagnosed by imaging (a lesion that has received local treatment needs to show clear progression to be considered a measurable lesion);

5.Expected survival time ≥ 12 weeks;

6.Normal function of major organs;

7.The subject voluntarily participates in this study, signs the informed consent form, has good compliance, and cooperates with the follow-up.

Exclusion Criteria:

1. Known or suspected to have a severe allergic history to the drugs related to this study (including drugs of the same type);
2. Evidence of liver decompensation: including but not limited to symptomatic ascites, esophageal-gastric variceal bleeding, hepatic encephalopathy, hepatorenaHave central nervous system metastasis;l syndrome, sepsis, etc.;
3. Have central nervous system metastasis;
4. Have a history of organ transplantation or are preparing for organ transplantation (including but not limited to liver transplantation);
5. Have a history of abdominal wall fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months before the start of treatment in the study;
6. Other situations in which the investigator deems that the subject should not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by RECIST V1.1 | up 2 years
  The ORR is defined as complete remission (CR) rate + partial remission (PR) rate by RECIST V1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by mRECIST | up 2 years
  The ORR is defined as complete remission (CR) rate + partial remission (PR) rate by mRECIST.
Disease control rate (DCR) by RECIST V1.1 | up 2 years
  The DCR is defined as complete remission (CR) rate + partial remission (PR) rate + stable disease (SD).
Progression-free survival (PFS) | up 2 years
  The PFS is defined as Time from the date of enrollment to of disease.
Overall survival (OS) | up 2 years
  The OS is defined as time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No